CLINICAL TRIAL: NCT05447377
Title: A Phase III, Multicenter, Double Blind, Randomized Study of SII Yellow Fever Vaccine to Compare Safety and Immunogenicity With STAMARIL® In Healthy Infants
Brief Title: A Study of SII Yellow Fever Vaccine to Compare Safety and Immunogenicity With STAMARIL® In Healthy Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YWF:02
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SII Yellow Fever Vaccine Lot A (Experimental): SII-YFV Lot A:
  SII Yellow Fever vaccine is Live attenuated Yellow Fever Virus (17D-213 Strain) not less than 1000 IU/dose propagated in specific pathogen-free chick embryos.
  Diluent: 0.5 mL of sterile water for injection
  In this arm a total of 554 participants will be enrolled. All participants will receive a single dose of SII-YFV Lot A will be administered concomitantly with an MMR and a Men A vaccine.
  Interventions: Biological: SII Yellow Fever Vaccine
- SII Yellow Fever Vaccine Lot B (Experimental): SII-YFV Lot B:
  SII Yellow Fever vaccine is Live attenuated Yellow Fever Virus (17D-213 Strain) not less than 1000 IU/dose propagated in specific pathogen-free chick embryos.
  Diluent: 0.5 mL of sterile water for injection
  In this arm a total of 554 participants will be enrolled. All participants will receive a single dose of SII-YFV Lot B will be administered concomitantly with an MMR and a Men A vaccine.
  Interventions: Biological: SII Yellow Fever Vaccine
- SII Yellow Fever Vaccine Lot C (Experimental): SII-YFV Lot C:
  SII Yellow Fever vaccine is Live attenuated Yellow Fever Virus (17D-213 Strain) not less than 1000 IU/dose propagated in specific pathogen-free chick embryos.
  Diluent: 0.5 mL of sterile water for injection
  In this arm a total of 554 participants will be enrolled. All participants will receive a single dose of SII-YFV Lot C will be administered concomitantly with an MMR and a Men A vaccine.
  Interventions: Biological: SII Yellow Fever Vaccine
- STAMARIL® (Active Comparator): STAMARIL is a Live attenuated Yellow Fever Virus (17D-204 Strain) not less than 1000 IU/dose produced in specified pathogen-free chick embryos.
  Solvent: Sodium Chloride 2.0 mg; Water for injections up to 0.5 mL.
  In this arm a total of 554 participants will be enrolled. All participants will receive a single dose of STAMARIL will be administered concomitantly with an MMR and a Men A vaccine.
  Interventions: Biological: STAMARIL®

INTERVENTIONS:
Biological: SII Yellow Fever Vaccine — SII YF vaccine:
  Live attenuated Yellow Fever Virus (17D-213 Strain) not less than 1000 IU/dose propagated in specific pathogen-free chick embryos.
  SII-YFV contains the 17D-213 vaccine strain, a derivative of 17D-204 strain which is used in many currently produced yellow fever vaccines. SIIPL imported the YF WHO Primary Seed Virus lot 213-77 from National Institute for Biological Standards and Control (NIBSC) for preparation of the master seed virus, working seed virus and the vaccine.
  After reconstitution, 1 dose (0.5 mL) contains:
  * Yellow fever virus 17D-213 strain (live, attenuated) not less than 1000 IU propagated in specific pathogen-free chick embryos
  * Excipients with known effects:
  * This product contains approximately 5 mg of sorbitol per dose.
  Arms: SII Yellow Fever Vaccine Lot A; SII Yellow Fever Vaccine Lot B; SII Yellow Fever Vaccine Lot C
Biological: STAMARIL® — STAMARIL® contains the 17D-204 vaccine strain, which is used in many currently produced yellow fever vaccines. STAMARIL® is specific pathogen free embryonated hen's egg based and is prepared by harvesting and stabilizing the virus collected from the homogenized chicken embryos infected with YF vaccine virus.
  STAMARIL® will be used as a comparator in the study. It is a live, attenuated, freeze-dried (lyophilized) vaccine and is to be reconstituted with solvent.
  After reconstitution, 1 dose (0.5 mL) contains:
  * Yellow fever virus 17D-204 strain (live, attenuated) not less than 1000 IU propagated in specific pathogen-free chick embryos
  * Excipients with known effects:
  * This product contains approximately 8 mg of sorbitol (E420) per dose.
  Arms: STAMARIL®

SUMMARY:
The study is designed as a Phase III, double-blind, multi-center, randomized, active-controlled study in which four groups of participants (n=554 per group) will receive either one of three different manufacturing lots of SII-YFV or STAMARIL® - a licensed and WHO pre-qualified YFV.

DETAILED DESCRIPTION:
The study is designed as a Phase III, double-blind, multi-center, randomized, active-controlled study in which four groups of participants (n=554 per group) will receive either one of three different manufacturing lots of SII-YFV or STAMARIL® - a licensed and WHO pre-qualified YFV.

A single dose of either SII-YFV or STAMARIL® will be administered concomitantly with an MMR and a Men A vaccine. The study will start only after the approval from the applicable ethics committees and national regulatory agencies. Following parental / guardian consent, participants will be screened for eligibility based on the defined inclusion and exclusion criteria for the trial. There will be three scheduled visits during the study. A screening and vaccination visit (Day 0) followed by additional study visits on Day 28 and on Day 180 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants as established by medical history and clinical examination
2. Male or female infants aged 9 to < 12 months (from the day they reach 9 months-of-age until the day before they reach 12-months/1-year-of-age)
3. Parental/ guardian ability and willingness to provide informed consent (as per local requirements/procedures), and to adhere to the protocol requirements.
4. Intend to remain residing in the study area throughout study participation
5. Parents/guardians willing to avoid the use of traditional/herbal local medications and treatments in infants for the duration of the study

Exclusion Criteria:

1. Fever (> 37.5°C) or any clinically significant acute infection at time of vaccination [Temporary exclusion criteria - participants may be rescreened at least 48 hours after the last recorded fever].
2. Previous history of laboratory confirmed infection with yellow fever, measles, mumps, rubella, Neisseria meningitidis serogroup A, and other flaviviruses e.g., dengue fever, tick-borne-encephalitis (TBE), Japanese encephalitis (JE), West Nile virus (WNV), zika virus, etc.

5. Previous vaccination against yellow fever, measles, mumps, rubella, Neisseria meningitidis serogroup A, TBE, JE, or dengue fever.

6. Receipt of any vaccine within past 28 days or planned vaccination until completion of day 28 study visit 7. A known hypersensitivity to any of the vaccine components (including gelatin, eggs, egg products, or chicken protein) or history of a life threatening reaction to any past vaccine 8. Receipt of immunoglobulin therapy and/or blood products since birth or planned administration until completion of Day 28 visit 9. Current or planned participation in another interventional study at any point throughout the entire study period 10. Receipt of any other investigational product or unlicensed medication in the preceding 28 days, or planned use until completion of Day 28 visit 7. Presence of significant malnutrition (weight-for-height z-score < -3SD)

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2216 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
YF neutralizing antibody (NAb) seroconversion | Day 28 post-vaccination
  Non-inferiority of the immune responses generated by SII-YFV compared to STAMARIL® in terms of YF neutralizing antibody (NAb) seroconversion rates as determined by plaque reduction neutralization test (PRNT50).
  Percentage seroconversion* on Day 28 post-vaccination
  * Seroconversion is defined as a four-fold rise in YF NAb (PRNT50) titres from baseline

SECONDARY OUTCOMES:
Yellow Fever Vaccine GMTs | Day 0 pre-vaccination and Day 28 post-vaccination
  GMTs on Day 0 pre-vaccination and Day 28 post-vaccination
  Equivalence of the immune responses generated by three different manufacturing lots of SII-YFV

CONTACTS AND LOCATIONS:
Locations (2):
- Center for Vaccine Development, Bamako, Mali
- MRC Unit The Gambia at LSHTM, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this study will be made available upon publication to members of the scientific and medical community for non-commercial use only, upon email request to the corresponding author. other study details are available on clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of publication of the study data
Access Criteria: Local regulatory authorities, ethics committee